CLINICAL TRIAL: NCT03436043
Title: Does Transmural Plastic Stenting Prevent the Recurrence of Pancreatic Fluid Collection After Metal Stent Removal in Walled Off Necrosis With Disconnected Pancreatic Duct Syndrome ? -Prospective Randomized Controlled Trial
Brief Title: Impact of Transmural Plastic Stent on Recurrence of Pancreatic Fluid Collection After Metal Stent Removal in Disconnected Pancreatic Duct
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Principal Investigator, Mohan Ramchandani, Consultant Gastroenterologist, Asian Institute of Gastroenterology, India
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AIG-006
Record Dates: First submitted 2018-02-10; First posted 2018-02-19 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2018-02

CONDITIONS: Acute Pancreatitis Necrotizing
Keywords: Walled of necrosis
MeSH Terms: conditions — Pancreatitis, Acute Necrotizing

STUDY DESIGN:
Who Masked: Participant
Masking Description: single blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transmural stenting (Experimental): In patients of walled off necrosis with disconnected pancreatic duct syndrome, metal stent will be removed at 3-4 weeks followed by transmural plastic stenting in the residual cavity.
  Interventions: Device: Transmural Plastic stenting
- No stenting (No Intervention): In patients of walled off necrosis with disconnected pancreatic duct syndrome, metal stent will be removed at 3-4 weeks without any further intervention.

INTERVENTIONS:
Device: Transmural Plastic stenting — After metal stent removal in patients of disconnected pancreatic duct syndrome, transmural plastic- double pig tail stent will be placed into the residual necrotic cavity with the standard duodenoscope.
  Arms: Transmural stenting

SUMMARY:
Walled of necrosis (WON) is severe local complication of acute necrotizing pancreatitis. Disconnected pancreatic duct syndrome(DPDS) is commonly seen (50-60%) after necrotizing pancreatitis and has long term implication like recurrent pancreatic fluid collections (PFC)] requiring re-intervention. Incidence of recurrent PFC is more common in patients with DPDS (17-50%) compared to others. Studies has shown permanent in-dwelling transmural stent reduces recurrence of PFC (1.7% vs 17.4%, p<0.001). Nowadays,WON is effectively managed with endoscopic step up approach (96%). Several studies showed dedicated self-expandable metal stent (SEMS) are effective compared to the plastic stents in management of WON with decreased need of re-intervention. However, SEMS cannot be kept for longer duration because of associated adverse events. So, experts recommend to remove SEMS within 4-6 weeks of placement. Considering this background, study is planned with aim to see the effect of transmural plastic stenting on recurrence of PFC after SEMS removal in walled off necrosis with DPDS.

DETAILED DESCRIPTION:
Acute necrotizing pancreatitis (ANP) is lethal complication and account for 10-20% of total pancreatitis. Necrotic collection is seen in majority of ANP and >50% of necrotic collection transform into Walled of necrosis (WON). Management of WON is challenging and under progressive evolution. With the advent of "step up approach" WON is effectively managed with greater success. Various studies and meta-analysis proved the efficacy of dedicated self-expandable metal stents (SEMS) over plastic stent in WON management. Disconnected pancreatic duct syndrome (DPDS) is late complication of necrotizing pancreatitis and increasingly identified after necrosectomy. DPDS is defined as complete disruption of the main pancreatic duct, resulting in a variable portion of the upstream pancreatic gland becoming isolated from the main pancreatic duct downstream. Ductal disruption leads to accumulation of pancreatic juice forming pancreatic or peri-pancreatic fluid collection. Incidence of recurrence of PFC in DPD is ~ 50%. DPDS is a separate clinical entity which demands special strategic approach and requires frequent re-intervention (surgical/endoscopic). Treatment option for DPDS is controversial and not yet clearly defined. Studies have shown that long term transmural plastic stent placement can reduce the recurrence rate (Stent removed-17% vs stent left behind-1.7%). So, some experts recommend that transmural stents can be left in situ indefinitely to decrease recurrence of PFC. Nowadays, SEMS are widely used for management of WON. However, metal stents cannot be kept for longer period because of increasing adverse events associated with longer duration (impaction/burring of SEMS in gastric wall, bleeding). So, recommendation is to remove SEMS as early as possible (within 4-6 weeks of drainage). Considering this fact, study is planned to evaluate the effect of transmural plastic stenting on recurrence of PFC after SEMS removal in walled off necrosis with DPDS. This will be randomised control study in patients with WON with DPDS who underwent SEMS drainage. After removal of SEMS patients with documented DPDS (magnetic resonance pancreatography and endoscopic retrograde pancreatography) will be randomised into 2 arms. In study arm after SEMS removal transmural plastic stent will be placed in to the cavity and in control arm SEMS will be removed with no transmural stenting. Thereafter patients will be followed at 3 months,6 months and yearly.

ELIGIBILITY:
Inclusion Criteria:

* All the patient who underwent EUS guided drainage with metal stent DPDS on MRCP & ERCP

Exclusion Criteria:

* Unwillingness to give written informed consent MRCP/ERCP-PD stricture ? (mimics DPD), leak Bleeding diathesis (Coagulopathy & thrombocytopenia) chronic pancreatitis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2017-10-20 (Actual); Primary Completion 2020-03-27 (Actual); Study Completion 2020-11-05 (Actual)

PRIMARY OUTCOMES:
Recurrence of PFC | 3 months
  In the study will see the re-ccurence of fluid collection in control and study arm

SECONDARY OUTCOMES:
Technical Success | 24 Months
  complication associated with deployment of transmural plastic, stent migration,recurrence of pancreatic fluid collection at 6 months and 1 year,new onset diabetes mellitus

CONTACTS AND LOCATIONS:
Locations (1):
- Asian Institute of Gastroenterology, Hyderabad, Andhra Pradesh, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chavan R, Nabi Z, Lakhtakia S, Gupta R, Jahangeer B, Talukdar R, Singh AP, Karyampudi A, Yarlagadda R, Ramchandani M, Kalapala R, Jagtap N, Reddy M, Tandan M, Rao GV, Reddy ND. Impact of transmural plastic stent on recurrence of pancreatic fluid collection after metal stent removal in disconnected pancreatic duct: a randomized controlled trial. Endoscopy. 2022 Sep;54(9):861-868. doi: 10.1055/a-1747-3283. Epub 2022 Feb 18. PMID 35180798